CLINICAL TRIAL: NCT05264636
Title: The Impact of a 28-day Steviol Glycoside Beverage on Human Gut Microflora Profile and Function vs. a Sucrose Beverage in Healthy Adults
Brief Title: The Impact of Steviol Glycosides on Human Gut Microflora Profile and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: INQ-2125
Record Dates: First submitted 2022-01-31; First posted 2022-03-03 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Healthy; Human Gut Microflora
Keywords: Steviol glycosides; gut microflora
MeSH Terms: interventions — Sucrose; Sugars; stevioside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: intervention products are coded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrose (Active Comparator): sucrose sweetened beverage 16 oz (473 ml) given daily for 28 days
  Interventions: Other: Sucrose
- Steviol glycosides (Experimental): steviol glycosides sweetened beverage 16 oz (473 ml) given daily for 28 days
  Interventions: Other: Steviol Glycosides

INTERVENTIONS:
Other: Sucrose — Sucrose Beverage
  Other Names: Sugar
  Arms: Sucrose
Other: Steviol Glycosides — Steviol Glycoside Beverage
  Other Names: Stevia
  Arms: Steviol glycosides

SUMMARY:
Diet and dietary ingredients can have a profound effect on gut microflora, both positive and negative. The reported effects on low and non caloric sweeteners (LNCS) on human gut microflora are contradictory in some of the in vitro and rodent studies. More specifically, the latter studies, using doses above the acceptable daily intake (ADI), suggest that LNCS may have adverse effects on gut microflora whereas recent data from human RCTs, using doses at or below the ADI, show little to no effect. In this study we will compare the effects of a low energy beverage made with steviol glycosides vs. a beverage made with sucrose on human gut microflora profile and function in a double blind, randomized study. A sucrose beverage was chosen as a control as it represents a caloric sugar sweetened beverage which is commonly consumed.

DETAILED DESCRIPTION:
This is a double blind randomized parallel study with 2 treatments to understand the effects of a low energy steviol glycoside beverage vs. a sucrose sweetened beverage on gut microflora profile and function over 28 days.

Participants will have a daily exposure to each test product for 28 days. (1) steviol glycosides (flavored water, steviol glycosides) and (2) sucrose (flavored water, sucrose). Individuals will be supplied with fecal collection kits to collect stool samples. The volunteers will be advised to collect a fecal sample before week 0(baseline), week 4(study end) and week 8(follow up period). Fecal microbial alpha diversity, beta diversity, and abundance of microbial taxa between the steviol glycoside and sucrose beverage consuming groups will be evaluated as well as fecal SCFA concentration, fasting serum insulin, glucose and lipids, weight, BMI, pulse and blood pressure at weeks 0(baseline),4(study end) and 8(follow up).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Non-pregnant, non-lactating individuals at least 25 of whom are male and 25 female
* Aged 18-50 years, inclusive
* BMI 18.5 to 24.9, inclusive
* Has access to a phone or tablet and wifi (to complete app based 3DDR)
* Consumption of ≤600ml (20oz) high intensity sweetened beverages per week for 1 month before screening
* Normal bowel frequency (≥3 per week)
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study Principal investigator
* Willing to not significantly alter their normal diet, physical activity routine, fiber intake or consume prebiotics or probiotics during the 8-week treatment period.
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Use of prebiotic or probiotic supplement one month prior to the study and during the entire duration of the study
* Smokers (cigarettes, vape or marijuana)
* Habitual consumption of >1.5L sugar sweetened beverages (eg. juice, soft drinks) per day
* High alcohol consumption (>14 drinks per week and >4 drinks per day for males; and >7 drinks per week and >3 drinks per day for females), or history of alcohol abuse. Alcohol intake during the study must stay below these limits listed above
* History of major trauma or major medical or surgical event requiring hospitalization within 3 months of screening
* Individuals with diabetes, bariatric surgery, celiac disease, phenylketonuria, inflammatory bowel disease, moderate or severe renal failure, moderate or severe liver disease or any other medical conditions or medications that increase risk to the subject or others or may affect the results, as judged by the Principal Investigator
* Use of antibiotics within 3 months of screening or with a condition likely to require the use of antibiotics during the study
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test beverages.
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification.
* Reported weight change of > 5kg in the preceding 3 months
* Employed by the study sponsor or affiliated organizations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
The effects of daily steviol glycosides consumption compared to the effects of daily sucrose consumption over 28 days on the alpha diversity, beta diversity, and abundance of microbial taxa in the human gut of healthy adults. | 28 days
  shotgun metagenomic sequencing at baseline and after 28 day intervention

SECONDARY OUTCOMES:
The effects of a daily steviol glycoside beverages compared to a sucrose beverage on fecal microflora short chain fatty acid (SCFA) production over 28 days. | 28 days
  ultra-high performance liquid chromatography-tandem mass spectrometry (UPLC-MS/MS)
The effects of a daily steviol glycoside beverage compared to a sucrose beverage on body weight over 28 days | 28 days
  Weight is measured in kg by a digital weighing scale at baseline and at 28 days
The effects of a daily steviol glycoside beverage compared to a sucrose beverage on BMI over 28 days | 28 days
  BMI will be measured as kg/m^2 at baseline and at 28 days. Weight (in kg) and height (in meters) will be combined to report BMI
The effects of a daily steviol glycoside compared to a sucrose beverage on blood pressure over 28 days | 28 days
  Blood pressure (systolic and diastolic) will be measured as mmHg at baseline and at 28 days
The effects of a daily steviol glycoside beverage compared to a sucrose beverages on pulse over 28 days | 28 days
  pulse rate (BPM) will be measured over 30 seconds at baseline and at 28 days
The effects of a daily steviol glycoside beverage compared to a sucrose beverage on fasting blood insulin over 28 days | 28 days
  Fasting blood insulin mciU/dl at baseline and at 28 days
The effects of a daily steviol glycoside beverage compared to a sucrose beverage on fasting blood glucose over 28 days | 28 days
  Fasting blood glucose will be measured in mg/dl at baseline and at 28 days
The effects of a daily steviol glycoside beverage compared to a sucrose beverage on fasting blood lipids over 28 days | 28 days
  Fasting blood lipids (total cholesterol, HDL, LDL, triglycerides) in mg/dl at baseline and at 28 days
Measurement and comparison of fecal microflora alpha diversity, beta diversity, and abundance of microbial taxa in the human gut of healthy adults at 28 days post intervention | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside or sucrose beverages. Microbial comparisons will be made by shotgun metagenomic sequencing on fecal samples taken at 28 days post intervention
The effects of a daily steviol glycoside beverage compared to a sucrose beverage on fecal short chain fatty acid (SCFA) production at 28 days post intervention | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside or sucrose beverage. Fecal SCFA production will be measured by ultra-high performance liquid chromatography-tandem mass spectrometry (UPLC-MS/MS) in fecal samples taken at 28 days post intervention
28 day post intervention changes in body weight | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. Body Weight will be measured in kg by a digital weighing scale at 28 days post intervention
28 day post intervention changes in BMI | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. BMI will be measured as kg/m^2 taken at 28 days post intervention. Weight (in kg) and height (in meters) will be combined to report BMI
28 day post intervention changes in Blood Pressure | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. Blood pressure (systolic and diastolic) will be measured as mmHg at 28 days post intervention
28 day post intervention changes in pulse rate | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. Pulse rate (BPM) will be measured over 30 seconds at 28 days post intervention
28 day post intervention changes in fasting blood insulin | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. Fasting blood insulin in mciU/dl taken at 28 days post intervention
28 day post intervention changes in fasting blood glucose | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. Fasting blood glucose will be measured in mg/dl taken at 28 days post intervention
28 day post intervention changes in fasting blood lipids | 28 days post intervention
  During a 28 day post intervention period, volunteers will not consume a steviol glycoside beverage or sucrose beverage. Fasting blood lipids (total cholesterol, HDL, LDL, triglycerides) in mg/dl taken at 28 days post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Inquis, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kwok D, Scott C, Strom N, Au-Yeung F, Lam C, Chakrabarti A, Hutton T, Wolever TM. Comparison of a Daily Steviol Glycoside Beverage compared with a Sucrose Beverage for Four Weeks on Gut Microbiome in Healthy Adults. J Nutr. 2024 Apr;154(4):1298-1308. doi: 10.1016/j.tjnut.2024.01.032. Epub 2024 Feb 24. PMID 38408729